CLINICAL TRIAL: NCT07153757
Title: A Prospective, Randomized, Open-label, Non-inferiority, Phase III Study Evaluating the Efficacy and Safety of 2 to 3 Years of Adjuvant Endocrine De-escalation Therapy for ER-positive/HER2-negative Stage I Breast Cancer
Brief Title: De-escalation Therapy in Stage I ER-Positive Breast Cancer: A Non-Inferiority Trial
Acronym: DESCENT
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Zhimin Shao, Professor, Fudan University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SCHBCC-N097
Record Dates: First submitted 2025-08-26; First posted 2025-09-04 (Actual); Last update posted 2025-09-04 (Actual); Status verified 2025-09

CONDITIONS: Breast Cancer Early Stage Breast Cancer (Stage 1-3)

STUDY DESIGN:
Intervention Model Description: Arm#1: 5 years of standard endocrine therapy； Arm#2: 2-3 years of de-escalated endocrine therapy
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 5 years of standard endocrine therapy (Active Comparator): The control group receives 5 years of standard endocrine therapy:
  Premenopausal patients: Tamoxifen (10 mg, orally, twice daily, for 5 years) or Toremifene (60 mg, orally, once daily, for 5 years); Postmenopausal patients: Letrozole (2.5 mg, orally, once daily, for 5 years) or Anastrozole (1 mg, orally, once daily, for 5 years) or Exemestane (25 mg, orally, once daily, for 5 years); A sequential regimen of 2-3 years of Tamoxifen or Toremifene followed by 3-2 years of Letrozole, Anastrozole, or Exemestane is acceptable.
  Ovarian function suppression is permitted for premenopausal patients. CDK4/6 inhibitors are not allowed during the treatment course
  Interventions: Drug: Endocrine Therapy of Physician's Choice
- 2-3 years of de-escalated endocrine therapy (Experimental): The experimental group receives 2-3 years of endocrine therapy:
  Premenopausal patients: Tamoxifen (10 mg, orally, twice daily, for 2-3 years) or Toremifene (60 mg, orally, once daily, for 2-3 years); Postmenopausal patients: Letrozole (2.5 mg, orally, once daily, for 2-3 years) or Anastrozole (1 mg, orally, once daily, for 2-3 years) or Exemestane (25 mg, orally, once daily, for 2-3 years).
  Ovarian function suppression is permitted for premenopausal patients. CDK4/6 inhibitors are not allowed during the treatment course.
  Interventions: Drug: Endocrine Therapy of Physician's Choice

INTERVENTIONS:
Drug: Endocrine Therapy of Physician's Choice — This study employs a 2-3 year de-escalated endocrine therapy regimen in the experimental group, which distinguishes it from other escalation therapy studies.

SUMMARY:
This study is a prospective, randomized, open-label, non-inferiority Phase III clinical trial, planning to enroll 2,934 patients, with a 1:1 allocation to either the conventional endocrine therapy group or the de-escalation therapy group. The aim is to evaluate the safety and efficacy of 2-3 years of de-escalated endocrine therapy in patients with T1N0M0 potentially low-risk breast cancer, respectively.

ELIGIBILITY:
Inclusion Criteria:

* Females aged 18 years or older;
* Postoperative pathological stage I early breast cancer: histologically confirmed invasive carcinoma with a maximum diameter ≤2 cm and node-negative (N0);
* Immunohistochemistry (IHC) shows ER-positive (ER ≥50%), HER2 IHC score of 0, 1+, or 2+ with no amplification confirmed by FISH, and Ki-67 ≤20%;
* Presence of at least one of the following potential low-risk factors:

  1）Tumor size ≤1 cm, 2）21-gene recurrence score <11, 3）Fudan digital pathological subtype classified as SNF1, 4）Age ≥65 years;
* ECOG performance status of 0 or 1;
* Patients with bilateral synchronous invasive lesions are eligible if both lesions are ER-positive, HER2-negative, and meet the tumor size criteria;
* Normal major organ function, meeting the following criteria:

  1. Hematological: HB ≥90 g/L (no transfusion within 14 days), ANC ≥1.5×10⁹/L, PLT ≥100×10⁹/L;
  2. Biochemical: TBIL ≤1.5×ULN, ALT and AST ≤3×ULN, serum Cr ≤1×ULN, and creatinine clearance >50 mL/min (Cockcroft-Gault formula);
* Participants voluntarily enroll, sign informed consent, demonstrate good compliance, and cooperate with follow-up.

Exclusion Criteria:

* Primary tumor size >2 cm in maximum diameter and/or axillary lymph node positivity;
* Prior neoadjuvant therapy, any systemic therapy, or local therapy (except surgery), including chemotherapy, targeted therapy, radiotherapy, or endocrine therapy;
* Prior adjuvant chemotherapy;
* Use of CDK4/6 inhibitors in the adjuvant setting;
* History of other malignancies (except cured basal cell carcinoma or cervical carcinoma in situ);
* Metastasis at any site;
* Pregnancy, lactation, or women of childbearing potential unable to use effective contraception;
* Concurrent participation in other clinical trials;
* Severe cardiac, pulmonary, hepatic, or renal dysfunction; LVEF <50% (by echocardiography); severe cardio-cerebrovascular diseases within 6 months (e.g., unstable angina, chronic heart failure, uncontrolled hypertension >150/90 mmHg, myocardial infarction, or stroke); poorly controlled diabetes; severe hypertension;
* Severe or uncontrolled infections;
* History of drug abuse or psychiatric disorders;
* Patients deemed unsuitable for the study by the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2934 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2033-09-01 (Estimated); Study Completion 2033-09-01 (Estimated)

PRIMARY OUTCOMES:
5-year disease-free survival in the per-protocol population | 5 year
  The proportion of patients in a clinical trial who remained free of disease recurrence, secondary primary cancers, and death from the disease for five years following treatment initiation, calculated specifically among those who completed the study intervention as predefined in the trial protocol(i.e., without major deviations such as incomplete treatment, use of prohibited therapies, or significant protocol violations).

SECONDARY OUTCOMES:
5-year disease-free survival in the Full Analysis Set | 5 year
  The proportion of patients in a clinical trial who remained free of disease recurrence, secondary primary cancers, and death from the disease for five years after randomization or initiation of treatment, analyzed within the Full Analysis Set (FAS) population-which includes all subjects randomized (or initially assigned to a treatment group) following the intention-to-treat (ITT) principle, regardless of whether they fully received, discontinued, or deviated from the protocol.
5-year invasive breast cancer-free survival in the per-protocol population | 5 year
  The proportion of participants in a clinical trial who, after receiving the full intended course of treatment without major protocol deviations, remained free of invasive ipsilateral or contralateral breast cancer recurrence, distant metastatic invasive breast cancer, and death from any cause for a period of five years from the start of treatment or randomization.
Overall survival in the per-protocol population | 5 year
  The length of time from randomization or initiation of treatment until death from any cause, measured specifically among participants who completed the study intervention without major protocol deviations, such as insufficient treatment exposure, use of prohibited therapies, or significant violations of inclusion/exclusion criteria.
Quality of Life score in the per-protocol population | 5 year
  The quality of life of patients was assessed using the EORTC QLQ-C30 questionnaire before, during, and after treatment.
safety | 5 year
  the evaluation of the adverse effects and potential risks of an investigational medical product (e.g., drug, device, or intervention) on participants throughout the study.

CONTACTS AND LOCATIONS:
Locations (1):
- 270 Dongan Road, Fudan University Shanghai Cancer Center, Shanghai, China

IPD SHARING:
Plan to Share IPD: No